CLINICAL TRIAL: NCT01072357
Title: Safety and Efficacy of Bevacizumab in High-Risk Corneal Transplant Survival
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Reza Dana, MD (Other)
Responsible Party: Sponsor-Investigator, Reza Dana, MD, Principal Investigator, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-07-062
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Corneal Neovascularization; Corneal Graft Failure
Keywords: High-Risk Corneal Transplantation; Penetrating Keratoplasty; Neovascularization; Corneal Blood Vessels; Avastin; Bevacizumab; Corneal Graft
MeSH Terms: conditions — Corneal Neovascularization; Neovascularization, Pathologic | interventions — Bevacizumab; Carboxymethylcellulose Sodium; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Avastin® (bevacizumab) (Active Comparator): Treatment will begin on Day 0, immediately upon the conclusion of the penetrating keratoplasty procedure with an injection of 0.1 milliliter (mL) (2.5 mg) bevacizumab. Starting Day 1 post-transplant surgery, subjects will begin treatment with topical bevacizumab (1% solution). Topical treatment will be self-administered 4 times a day for 4 weeks.
  The study treatments are to be given in addition to standard of care treatments. Also, all patients will follow a standard post-operative follow-up visit schedule.
  Interventions: Drug: Avastin® (bevacizumab)
- 0.9% NaCl & Refresh Liquigel (Placebo Comparator): Treatment will begin on Day 0, immediately upon the conclusion of the penetrating keratoplasty procedure with an injection of 0.1 mL 0.9% sodium chloride (NaCl). Starting Day 1 post-transplant surgery, subjects will begin treatment with topical Refresh Liquigel. Topical treatment will be self-administered 4 times a day for 4 weeks.
  The study treatments (both topical and subconjunctival injection) are to be given in addition to standard of care treatments. Also, all patients will follow a standard post-operative follow-up visit schedule.
  Interventions: Drug: 0.9% NaCl & Refresh Liquigel

INTERVENTIONS:
Drug: Avastin® (bevacizumab) — One time subconjunctival injection of 0.1 mL (2.5 mg) bevacizumab followed by topical treatment with 1% solution bevacizumab four times a day for four weeks.
  Other Names: Avastin; bevacizumab
  Arms: Avastin® (bevacizumab)
Drug: 0.9% NaCl & Refresh Liquigel — One-time subconjunctival injection of 0.1mL 0.9% NaCl followed by topical treatment with Refresh Liquigel four times a day for four weeks
  Other Names: Sodium Chloride; Refresh Liquigel; NaCL
  Arms: 0.9% NaCl & Refresh Liquigel

SUMMARY:
The leading risk factor for corneal transplant rejection is abnormal blood vessel growth of the host bed. Vascular endothelial growth factor (VEGF) is thought to be a mediator of this corneal neovascularization (NV), therefore we would like to test the safety and efficacy of local VEGF blockade in the promotion of graft survival in high risk corneal transplants.

DETAILED DESCRIPTION:
The purpose of this study is to test the effectiveness of a drug, bevacizumab (Avastin), in preventing blood vessels that often occur after a corneal transplantation which are considered at "high-risk" for rejection. In many cases these blood vessels lead to the graft rejection and eventual failure of the corneal transplant. It is hoped that this treatment will increase the chances of corneal graft survival.

The medication used in this study is called bevacizumab or Avastin (Genentech, Inc). It works by inhibiting the action of a molecule called vascular endothelial growth factor (VEGF). VEGF is a substance molecule that binds to certain cells to stimulate new blood vessel formation. When VEGF is bound to the drug, it cannot stimulate the formation and growth of new blood vessels. Growth of blood vessels into the cornea is a complication which can worsen the prognosis of your corneal transplant and put the transplant at a higher risk for rejection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient or legally authorized representative willing and able to provide written informed consent
* Willing and able to comply with study assessments for the full duration of the study
* High-risk characteristics for penetrating keratoplasty: Either presence of 1.) Corneal NV in one or more quadrants (≥ 3 clock hours NV ≥ 2mm from the limbus) OR 2.) Extension of corneal NV to graft-host junction in a previous failed graft
* In generally good stable overall health

Exclusion Criteria:

* History of Stevens-Johnson syndrome or ocular pemphigoid
* Ocular or periocular malignancy
* Non-healing epithelial defect of at least 0.5x0.5 mm in host corneal bed lasting ≥6 weeks preoperatively
* Uncontrolled glaucoma
* Currently on dialysis
* Has received treatment with anti-VEGF agents (intraocular or systemic) within 45 days of study entry
* Concurrent use of systemic anti-VEGF agents
* Change in topical corticosteroid regimen within 14 days of transplantation
* Use of systemic immunosuppressive for indication other than corneal graft rejection
* Pregnancy (positive pregnancy test) or lactating
* Pre-menopausal women not using adequate contraception (Reliable intrauterine devices, hormonal contraception or a spermicide in combination with a barrier method)
* Uncontrolled hypertension defined as systolic blood pressure (BP) ≥150 or diastolic BP ≥90 mmHg
* History of thromboembolic event within 12 months prior to study entry
* Participation in another simultaneous medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Dana, MD, MPH, MSc, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Avastin® (Bevacizumab): Treatment will begin on Day 0, immediately upon the conclusion of the penetrating keratoplasty procedure with an injection of 0.1 milliliter (mL) (2.5 mg) bevacizumab. Starting Day 1 post-transplant surgery, subjects will begin treatment with topical bevacizumab (1% solution). Topical treatment will be self-administered 4 times a day for 4 weeks.
  The study treatments are to be given in addition to standard of care treatments. Also, all patients will follow a standard post-operative follow-up visit schedule.
  Avastin® (bevacizumab): One time subconjunctival injection of 0.1 mL (2.5 mg) bevacizumab followed by topical treatment with 1% solution bevacizumab four times a day for four weeks.
- 0.9% NaCl & Refresh Liquigel: Treatment will begin on Day 0, immediately upon the conclusion of the penetrating keratoplasty procedure with an injection of 0.1 mL 0.9% sodium chloride (NaCl). Starting Day 1 post-transplant surgery, subjects will begin treatment with topical Refresh Liquigel. Topical treatment will be self-administered 4 times a day for 4 weeks.
  The study treatments (both topical and subconjunctival injection) are to be given in addition to standard of care treatments. Also, all patients will follow a standard post-operative follow-up visit schedule.
  0.9% NaCl & Refresh Liquigel: One-time subconjunctival injection of 0.1mL 0.9% NaCl followed by topical treatment with Refresh Liquigel four times a day for four weeks
Period: Overall Study
Arm/Group | Avastin® (Bevacizumab) | 0.9% NaCl & Refresh Liquigel
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Avastin® (Bevacizumab) | 0.9% NaCl & Refresh Liquigel | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (17.0) | 63.0 (13.0) | 67.2 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 10 | 18
  Hispanic | 2 | 1 | 3
  African American | 4 | 3 | 7
  Asian | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Graft Failure at Week 39 and 52
Description: Time from surgery to overall graft failure (regardless of cause). Graft failure was monitored throughout the entire study, but only the time points at which graft failure occurred are reported below.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Avastin® (Bevacizumab) | 0.9% NaCl & Refresh Liquigel
Number analyzed (Participants) | 15 | 14
Participants
  39 Week Time Point | 0 | 1
  52 Week Time Point | 1 | 1

2. Secondary Outcome: Endothelial Cell Density
Description: Endothelial Cell Density (Assessed at Weeks 26 & 52). Measure of the number of cells present within the endothelium that are responsible for providing the cornea with nourishment.
Time Frame: 52 Weeks
Measure: Mean (Standard Deviation); unit: Number of cells per millimeters squared
Arm/Group | Avastin® (Bevacizumab) | 0.9% NaCl & Refresh Liquigel
Number analyzed (Participants) | 15 | 14
Number of cells per millimeters squared
  Week 26 Time Point | 1814.25 (729.72) | 2249.83 (891.25)
  Week 52 Time Point | 1432.50 (696.61) | 1926.67 (948.03)

ADVERSE EVENTS:
Time Frame: 52 Weeks
Arm/Group | Avastin® (Bevacizumab) | 0.9% NaCl & Refresh Liquigel
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/15
Other Adverse Events (participants affected / at risk) | 13/15 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin® (Bevacizumab) (N=15) | 0.9% NaCl & Refresh Liquigel (N=15)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin® (Bevacizumab) (N=15) | 0.9% NaCl & Refresh Liquigel (N=15)
Foreign Body Sensation (Eye disorders) | 5 (5) | 4 (4)
Tearing (Eye disorders) | 6 (7) | 4 (5)
Blurry Vision (Eye disorders) | 5 (5) | 3 (3)
Ocular Pain (Eye disorders) | 6 (7) | 4 (4)
Photophobia (Eye disorders) | 4 (5) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes